CLINICAL TRIAL: NCT05591430
Title: Bilateral Pulsed Radiofrequency of Dorsal Root Ganglia of S2-4 Versus Ganglion Impar Neurolysis for Severe Perianal and Perineal Pain in Cancer Patients
Brief Title: Pulsed Radiofrequency of S2-4 Versus Ganglion Impar Neurolysis for Severe Perianal and Perineal Pain in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Walaa Youssef Elsabeeny, Assistant professor of Anesthesia and Pain management, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AP2207-50108
Record Dates: First submitted 2022-10-19; First posted 2022-10-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ganglion Impar Neurolysis (Active Comparator): Block of ganglion impar using neurolytic
  Interventions: Procedure: Ganglion Impar Neurolysis
- Bilateral S2, S3 and S4 Pulsed radiofrequency (Experimental): Pulsed radiofrequency of S2-S4
  Interventions: Procedure: Bilateral S2, S3 and S4 Pulsed radiofrequency

INTERVENTIONS:
Procedure: Ganglion Impar Neurolysis — block of Ganglion Impar by neurolytic drug
  Arms: Ganglion Impar Neurolysis
Procedure: Bilateral S2, S3 and S4 Pulsed radiofrequency — Bilateral S2, S3 and S4 Pulsed radiofrequency
  Arms: Bilateral S2, S3 and S4 Pulsed radiofrequency

SUMMARY:
Perineal pain resulting from malignancy is usually severe. Pain can be related to the malignancy or as a complication related to the treatment. several modalities are adopted to control such pain starting from medical management to interventional pain procedures.

DETAILED DESCRIPTION:
Perineal pain resulting from malignancy is usually severe. Pain can be related to the malignancy or as a complication related to the treatment. several modalities are adopted to control such pain starting from medical management to interventional pain procedures. Ganglion impar block has been traditionally used for treatment of such perineal pain. Radiofrequency of sacral dorsal root ganglia can be used as an alternative for pain control.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-75 years
* ASA II-III with perianal and perineal pain related to cancer

Exclusion Criteria:

* patient refusal
* coagulation defects
* abnormal kidney or liver functions
* local infection at site of injection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2024-05-25 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | 2 hours
  the score of visual analogue scale score, with minimum score of 0 and maximum of 10, with higher scores meaning more severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Walaa Y Elsabeeny, MD, Principal Investigator — Assistant professor of Anesthesia and Pain Management, National Cancer Institute, Cairo University
Locations (1):
- Walaa Y Elsabeeny, Cairo, Egypt